CLINICAL TRIAL: NCT00002566
Title: INTERNATIONAL RANDOMIZED STUDY FOR THE SALVAGE TREATMENT OF GERM CELL TUMOURS
Brief Title: Combination Chemotherapy With Bone Marrow Transplantation in Treating Men With Germ Cell Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000063579; FRE-IT94; FRE-FNCLCC-IT94; NCI-F94-0019
Record Dates: First submitted 1999-11-01; First posted 2004-01-15 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Extragonadal Germ Cell Tumor; Testicular Germ Cell Tumor
Keywords: recurrent malignant testicular germ cell tumor; extragonadal germ cell tumor
MeSH Terms: conditions — Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; Ifosfamide; Vinblastine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: ifosfamide
Drug: vinblastine sulfate
Procedure: autologous bone marrow transplantation
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not known whether combining chemotherapy with bone marrow transplantation is a more effective treatment for men with germ cell tumors.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with bone marrow transplantation in treating men with relapsed germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the event-free survival of male patients with germ cell tumors in relapse or first partial remission treated with salvage therapy comprising cisplatin, etoposide, and ifosfamide (PEI) or vinblastine, ifosfamide, and cisplatin (VeIP) with or without high-dose carboplatin, etoposide, and cyclophosphamide, followed by autologous bone marrow and/or peripheral blood stem cell transplantation.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior complete remission to first-line treatment (yes vs no), primary site of disease (testicular vs retroperitoneal vs mediastinal), and lung metastases at study entry (yes vs no). Autologous bone marrow and peripheral blood stem cells (PBSC) are harvested. Part I (salvage): Patients are assigned to regimen A if they previously received vinblastine as part of a first-line treatment, such as cisplatin, vinblastine, and bleomycin (PVB) or cisplatin, cyclophosphamide, doxorubicin, vinblastine, and bleomycin (CISCA VB). Patients are assigned to regimen B if they previously received etoposide (VP-16) as part of a first-line treatment, such as bleomycin, VP-16, and cisplatin (BEP). Regimen A: Patients receive cisplatin IV over 2 hours, VP-16 IV over 2 hours, and ifosfamide IV over 1 hour on days 1-5 (PEI). Regimen B: Patients receive cisplatin and etoposide as in regimen A and vinblastine IV on days 1 and 2 (VeIP). Treatment on both regimens continues every 3 weeks for 2 courses. Patients with refractory disease at day 43 are taken off study. Part II: Patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive 2 additional courses of PEI or VeIP. Arm II: Patients receive 1 additional course of PEI or VeIP, followed by 1 course of high-dose carboplatin IV over 2 hours, VP-16 IV over 2 hours, and cyclophosphamide IV over 1 hour on days 1-4. Autologous bone marrow and/or PBSC are reinfused on day 7 of the fourth course for patients on both arms. Patients on both arms with residual disease after the fourth course may undergo surgery.

PROJECTED ACCRUAL: A total of 280 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of testicular or extragonadal male germ cell tumors Must meet 1 of the following conditions after completion of platinum-based first-line chemotherapy: Complete remission (CR) followed by relapse Partial remission (PR) Prior resection of viable malignancy with elevated tumor markers allowed Initial bulky disease with no CR (significantly reduced but still abnormal in plateau) allowed if there is an increase in biological tumor markers or development of new metastases Seminoma with relapse after CR or PR to cisplatin-based chemotherapy allowed No pure seminoma pre-treated with carboplatin No refractory disease (i.e., documented increase in tumor burden and/or serum tumor marker level during or within 1 month after platinum-containing chemotherapy) CNS involvement allowed

PATIENT CHARACTERISTICS: Age: 16 and over Sex: Male Performance status: WHO 0-2 OR Karnofsky 50-100% Life expectancy: No limits on life expectancy due to severe non-malignant disease Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No severe cardiac disease that would interfere with study therapy Pulmonary: No severe pulmonary disease that would interfere with study therapy Other: HIV negative No severe neurologic or metabolic disease that would interfere with study therapy No psychological, socioeconomic, or geographic circumstances that would preclude study No other concurrent malignancy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy for metastatic disease allowed Surgery: See Disease Characteristics Prior surgery for metastatic disease allowed

Ages: 16 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 1994-02 (Actual); Primary Completion 2001-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Louis Pico, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France